CLINICAL TRIAL: NCT03137355
Title: The International Registry for Leigh Syndrome
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mary Kay Koenig, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-14-0907
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Leigh Syndrome; Leigh Disease; Leigh's Necrotizing Encephalopathy; Subacute Necrotizing Encephalomyopathy; Subacute Necrotizing Encephalomyelopathy
Keywords: Leigh Syndrome; Leigh Disease; Leigh's Necrotizing Encephalopathy; Subacute Necrotizing Encephalomyelopathy; Subacute Necrotizing Encephalomyopathy
MeSH Terms: conditions — Leigh Disease; Necrotizing encephalopathy, infantile subacute, of Leigh

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Leigh syndrome: All people diagnosed with Leigh syndrome.

SUMMARY:
The purpose of this study is to develop a database containing clinical and laboratory information for patients with Leigh syndrome. The goal is to provide a greater understanding of Leigh syndrome allowing further characterization of this disease.

DETAILED DESCRIPTION:
Leigh syndrome, also known as juvenile sub-acute necrotizing encephalopathy, is a progressive neurodegenerative disorder associated with dysfunction of mitochondrial oxidative phosphorylation (OXPHOS). First described in 1951 by British neuropsychiatrist Archibald Denis Leigh, the condition has evolved from a post mortem diagnosis to a clinical entity with characteristic radiologic and laboratory findings.

Leigh syndrome is a rare and heterogeneous disease, finding a substantial number of patients to study is difficult. The lack of natural history data in Leigh syndrome and the small number of patients included in clinical reports thus far has limited the ability to fully comprehend the progression of this disease and assess prognostic factors. A Leigh syndrome database will help improve our understanding of this rare disease leading to an improved ability to predict outcomes and/or improve treatment paradigms. Collecting natural history data on Leigh syndrome and integrating this information into a database will be useful in understanding the course of the disease and identifying trends.

ELIGIBILITY:
Inclusion Criteria:

* All participants with a diagnosis of Leigh syndrome will be invited to participate

Exclusion Criteria:

* People without Leigh syndrome

Ages: 0 Days to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with a diagnosis of Leigh syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06-17 (Actual); Primary Completion 2030-06-17 (Estimated); Study Completion 2030-06-17 (Estimated)

PRIMARY OUTCOMES:
Phenotypical characteristics of Leigh syndrome | 10 years
  The goal of this project is to collect longitudinal data on the natural history of Leigh syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Koenig, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- See also: Related Info — http://peopleagainstleighs.org/registry/